CLINICAL TRIAL: NCT02351479
Title: Hula, a Physical Activity Intervention for Female-Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Bantum-2013-2
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity; Breast Cancer; Cervical Cancer; Ovarian Cancer; Endometrial Cancer
Keywords: hula; breast cancer; female; hawaii; physical activity; cervical cancer; ovarian cancer; endometrial cancer
MeSH Terms: conditions — Motor Activity; Breast Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hula (Other): Hula is an ancient, Native Hawaiian dance form of cultural expression and physical activity. Participants will attend one-hour hula classes twice a week for six months.
  Interventions: Behavioral: Hula

INTERVENTIONS:
Behavioral: Hula

SUMMARY:
A six-month interventional program to determine the biological and psychosocial effects of hula as a form of physical activity for female breast, cervical, endometrial or ovarian cancer survivors living on Oahu.

ELIGIBILITY:
Inclusion Criteria:

* Lives on Oahu
* Diagnosed with primary breast,cervical, endometrial or ovarian cancer (stage I-III)
* Completed initial regional and systemic treatment for breast cancer 2 months ago
* Physically capable of doing the hula-based physical activity
* Receives approval by attending physician to participate in trial

Exclusion Criteria:

* Currently undergoing chemotherapy or radiation therapy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hula Program Feasibility (Compliance as measured by the proportion of total sessions attended and a questionnaire regarding satisfaction with the program at the end of the intervention) | 6 months after the start of the intervention program
  Compliance as measured by the proportion of total sessions attended and a questionnaire regarding satisfaction with the program at the end of the intervention

SECONDARY OUTCOMES:
Biomarkers - Sex Hormones (Circulating levels of sex hormones measured in serum samples) | Baseline, 6 months and 12 months after the start of the intervention program
  Circulating levels of sex hormones measured in serum samples.
Biomarkers - Cytokines (Circulating levels of cytokines measured in serum samples.) | Baseline, 6 months and 12 months after the start of the intervention program
  Circulating levels of cytokines measured in serum samples.
Biomarkers - Inflammatory Markers (Circulating levels of leptin, CRP, IGF-1, and IGFBP3 measured in serum samples collectively.) | Baseline, 6 months and 12 months after the start of the intervention program
  Circulating levels of leptin, CRP, IGF-1, and IGFBP3 measured in serum samples collectively.
DNA Methylation Patterns (DNA methylation patterns as detected with the Illumina Assay containing methylation sites in RefSeq genes and CpG islands collectively.) | Baseline, 6 months and 12 months after the start of the intervention program
  DNA methylation patterns as detected with the Illumina Assay containing methylation sites in RefSeq genes and CpG islands collectively.
Self-Report Outcomes - Demographics (Collectively looking at demographic items as measured on the baseline questionnaire, including ethnicity, education, family, history of cancer, stage of cancer, treatment type, and comorbidities.) | Baseline, 6 months and 12 months after the start of the intervention program
  Collectively looking at demographic items as measured on the baseline questionnaire, including ethnicity, education, family, history of cancer, stage of cancer, treatment type, and comorbidities.
Self-Report Outcomes - Physical Activity (Minutes per week of exercise assessed using The Women's Health Initiative Physical Activity Questionnaire) | Baseline, 6 months and 12 months after the start of the intervention program
  Minutes per week of exercise assessed using The Women's Health Initiative Physical Activity Questionnaire
Self-Report Outcomes - Health-Related Quality of Life (Quality of life of participants assessed using The European Organization for Research and Treatment of Cancer QLQ-C30.) | Baseline, 6 months and 12 months after the start of the intervention program
Self-Report Outcomes - Fatigue (assessed using The Brief Fatigue Inventory (BFI) | Baseline, 6 months and 12 months after the start of the intervention program
  The severity and impact of fatigue on daily functioning assessed using The Brief Fatigue Inventory (BFI).
Self-Report Outcomes - Depression (indicated using The Centers for Epidemiological Studies Depression Scale (CES-ED) | Baseline, 6 months and 12 months after the start of the intervention program
  The presence of depression as indicated using The Centers for Epidemiological Studies Depression Scale (CES-ED).
Self-Report Outcomes - Affective States (assessed using The Profile of Mood States short form (POMS-SF) questionnaire.) | Baseline, 6 months and 12 months after the start of the intervention program
  Affect of participants assessed using The Profile of Mood States short form (POMS-SF) questionnaire.
Self-Report Outcomes - Social Constraints (assessed using The 10-item Social Constraints Scale.) | Baseline, 6 months and 12 months after the start of the intervention program
  How people adjust and cope with a cancer diagnosis assessed using The 10-item Social Constraints Scale.
Self-Report Outcomes - Cognitive Functioning (assessed using the 42-item FACTcog | Baseline, 6 months and 12 months after the start of the intervention program
  2 subscales assess cognitive deficiency and cognitive capability

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bantum, MA, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bantum EO, Yamada PM, Makolo T, Yu H, Pagano I, Subia N, Walsh C, Loo LWM. Hula as a physical activity and social support intervention for sustained activity in female breast and gynecologic cancer survivors. Front Psychol. 2023 Oct 24;14:1190532. doi: 10.3389/fpsyg.2023.1190532. eCollection 2023. PMID 37941759